CLINICAL TRIAL: NCT00699608
Title: A Randomised, Double-blind, Double-dummy, Placebo-controlled, 3-way Crossover Study to Evaluate Potential Next-day Residual Effects of a Single Evening Dose of 3mg Eszopiclone and 7.5mg Zopiclone in Healthy Adult Subjects.
Brief Title: An Evaluation of Potential Next-day Residual Effects of Eszopiclone in Healthy Volunteers.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ESZ111503
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Results first posted 2010-05-12 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2011-03

CONDITIONS: Healthy Subjects; Sleep Initiation and Maintenance Disorders
Keywords: Zopiclone; Hypnotic; Residual effects; Eszopiclone
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — zopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Crossover (Experimental): All subjects received all three treatments in a randomised order
  Interventions: Drug: GSK1755165; placebo; zopiclone

INTERVENTIONS:
Drug: GSK1755165; placebo; zopiclone — Subjects receive either 3mg GSK1755165, matching placebo or 7.5mg zopiclone

SUMMARY:
This study will explore potential next-day residual effects of a single evening dose of 3mg of the hypnotic, eszopiclone, 7.5mg of zopiclone, and placebo, in healthy adult subjects.

ELIGIBILITY:
INCLUSION CRITERIA:

* Healthy male and female subjects providing written informed consent.

EXCLUSION CRITERIA:

* Significant medical disorders;
* Sleeping difficulties; alcohol and/or substance abuse;
* Recent use of psychotropic medications, or need to use them during study;
* Very high BMI or very low BMI or bodyweight;
* Known hypersensitivity to the study medications or their excipients;
* Unwilling or unable to meet certain lifestyle or dietary restrictions during the study.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2008-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Guildford, Surrey, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Eszopiclone First, Zopiclone Second, Placebo Third: 3 mg eszopiclone during first intervention period, 7.5 mg zopiclone during second intervention period (after 4-14 day washout period), placebo during third intervention period (after 4-14 day washout period)
- Eszopiclone First, Placebo Second, Zopiclone Third: 3 mg eszopiclone during first intervention period, placebo during second intervention period (after 4-14 day washout period), 7.5 mg zopiclone during third intervention period (after 4-14 day washout period)
- Zopiclone First, Eszopiclone Second, Placebo Third: 7.5 mg zopiclone during first intervention period, 3 mg eszopiclone during second intervention period (after 4-14 day washout period), placebo during third intervention period (after 4-14 day washout period)
- Zopiclone First, Placebo Second, Eszopiclone Third: 7.5 mg zopiclone during first intervention period, placebo during second intervention period (after 4-14 day washout period), 3 mg eszopiclone during third intervention period (after 4-14 day washout period)
- Placebo First, Eszopiclone Second, Zopiclone Third: Placebo during first intervention period, 3 mg eszopiclone during second intervention period (after 4-14 day washout period), 7.5 mg zopiclone during third intervention period (after 4-14 day washout period)
- Placebo First, Zopiclone Second, Eszopiclone Third: Placebo during first intervention period, 7.5 mg zopiclone during second intervention period (after 4-14 day washout period), 3 mg eszopiclone during third intervention period (after 4-14 day washout period)
Period: First Intervention
Arm/Group | Eszopiclone First, Zopiclone Second, Placebo Third | Eszopiclone First, Placebo Second, Zopiclone Third | Zopiclone First, Eszopiclone Second, Placebo Third | Zopiclone First, Placebo Second, Eszopiclone Third | Placebo First, Eszopiclone Second, Zopiclone Third | Placebo First, Zopiclone Second, Eszopiclone Third
Started | 16 | 15 | 15 | 15 | 15 | 15
Completed | 16 | 15 | 14 | 15 | 14 | 15
Not Completed | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0
Period: First 4-14 Day Washout Period
Arm/Group | Eszopiclone First, Zopiclone Second, Placebo Third | Eszopiclone First, Placebo Second, Zopiclone Third | Zopiclone First, Eszopiclone Second, Placebo Third | Zopiclone First, Placebo Second, Eszopiclone Third | Placebo First, Eszopiclone Second, Zopiclone Third | Placebo First, Zopiclone Second, Eszopiclone Third
Started | 16 | 15 | 14 | 15 | 14 | 15
Completed | 16 | 15 | 14 | 15 | 14 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Eszopiclone First, Zopiclone Second, Placebo Third | Eszopiclone First, Placebo Second, Zopiclone Third | Zopiclone First, Eszopiclone Second, Placebo Third | Zopiclone First, Placebo Second, Eszopiclone Third | Placebo First, Eszopiclone Second, Zopiclone Third | Placebo First, Zopiclone Second, Eszopiclone Third
Started | 16 | 15 | 14 | 15 | 14 | 15
Completed | 16 | 15 | 13 | 14 | 14 | 15
Not Completed | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Period: Second 4-14 Day Washout Period
Arm/Group | Eszopiclone First, Zopiclone Second, Placebo Third | Eszopiclone First, Placebo Second, Zopiclone Third | Zopiclone First, Eszopiclone Second, Placebo Third | Zopiclone First, Placebo Second, Eszopiclone Third | Placebo First, Eszopiclone Second, Zopiclone Third | Placebo First, Zopiclone Second, Eszopiclone Third
Started | 16 | 15 | 13 | 14 | 14 | 15
Completed | 16 | 15 | 13 | 14 | 14 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Eszopiclone First, Zopiclone Second, Placebo Third | Eszopiclone First, Placebo Second, Zopiclone Third | Zopiclone First, Eszopiclone Second, Placebo Third | Zopiclone First, Placebo Second, Eszopiclone Third | Placebo First, Eszopiclone Second, Zopiclone Third | Placebo First, Zopiclone Second, Eszopiclone Third
Started | 16 | 15 | 13 | 14 | 14 | 15
Completed | 16 | 15 | 13 | 14 | 14 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 91
Age Continuous [Mean (Standard Deviation); unit: years] | 29.8 (3.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 45
Race/Ethnicity, Customized [Number; unit: participants]
  White | 63
  African American/African Heritage | 14
  Asian-Central/South Asian Heritage | 6
  Asian-South East Asian Heritage | 5
  Asian-East Asian Heritage | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Tracking Error Assessed During the Continuous Tracking Test (CTT)
Description: Analysis was performed on the mean of the five assessments conducted 7.5, 8, 8.5, 9, and 9.5 hours post-dose (double-blind) The CTT is a task (duration of 8 minutes) of psychomotor function that entails using a slider to keep a cursor in alignment with a moving target on a visual display unit screen. The movement of the target is the function of an irregular sine wave, and cursor accuracy is measured by the mean tracking error - the difference between the centers of target and cursor in pixels, sampled 5 times per second, over the test. Lower scores are indicative of more accurate tracking.
Time Frame: 7.5, 8, 8.5, 9, and 9.5 hours post-dose (double-blind)
Population: Intent-to-Treat (ITT) Population: all subjects who gave informed consent, were randomised, and received at least one dose of double-blind medication. Only participants who had assessment of the measure the day after double-blind treatment were analyzed.
Measure: Least Squares Mean (Standard Error); unit: pixels
Groups:
- Placebo: Placebo
- Eszopiclone: 3 mg Eszopiclone
- Zopiclone: 7.5 mg Zopiclone
Arm/Group | Placebo | Eszopiclone | Zopiclone
Number analyzed (Participants) | 89 | 87 | 90
pixels | 10.29 (0.625) | 12.49 (0.634) | 13.48 (0.621)
Statistical Analysis 1: Comparison: Eszopiclone vs Zopiclone; Test type: Superiority or Other; p = 0.267, ANCOVA; ANCOVA used (fixed effects: adjusted period baseline, participant baseline, age, gender, period and treatment group; random effect: participant); Mean Difference (Final Values) = -0.99, 95% CI [-2.74 to 0.76]

2. Secondary Outcome: Mean Tracking Error (MTE) Assessed During the CTT
Description: Analysis was performed on the individual assessments conducted at 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind) . The CTT is a task (8 minute duration) of psychomotor function that entails using a slider to keep a cursor in alignment with a moving target on a visual display unit screen. The movement of the target is the function of an irregular sine wave, and cursor accuracy is measured by the MTE, the difference between the centers of target and cursor in pixels, sampled 5 times per second, over the test. Lower scores are indicative of more accurate tracking.
Time Frame: 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind)
Population: Intent-to-Treat (ITT) Population: all participants who gave informed consent, were randomised, and received at least one dose of double-blind study medication. Only participants who had assessment of the measure the day after double-blind treatment were analyzed.
Measure: Least Squares Mean (Standard Error); unit: pixels
Arm/Group | Placebo | Eszopiclone | Zopiclone
Number analyzed (Participants) | 89 | 87 | 90
pixels
  7.5 hours post-dose | 10.20 (0.596) | 12.80 (0.602) | 13.07 (0.592)
  8 hours post-dose | 9.70 (0.830) | 12.72 (0.840) | 13.15 (0.826)
  8.5 hours post-dose | 10.08 (0.917) | 12.54 (0.928) | 12.93 (0.913)
  9 hours post-dose | 11.02 (0.214) | 13.00 (1.229) | 14.81 (1.208)
  9.5 hours post-dose | 10.44 (1.108) | 13.50 (1.121) | 13.55 (1.101)
  10 hours post-dose | 10.12 (1.057) | 12.85 (1.069) | 12.53 (1.051)
  10.5 hours post-dose | 9.48 (0.757) | 11.38 (0.767) | 11.84 (0.753)
  11 hours post-dose | 10.55 (0.822) | 10.86 (0.833) | 11.65 (0.818)
  11.5 hours post-dose | 9.18 (0.523) | 10.06 (0.530) | 10.30 (0.521)

3. Secondary Outcome: CTT Mean Reaction Time
Description: Analysis was performed on the individual assessments conducted at 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind) A further outcome derived from the CTT is a peripheral awareness task where the participant responds to a stimulus presented in the periphery of vision, while simultaneously attending to the tracking test. The mean reaction time, in milliseconds, to these stimuli over the trial period is taken as the response measure for this component of the divided attention task. A lower mean reaction time is indicative of better peripheral awareness.
Time Frame: 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind)
Population: Intent-to-Treat (ITT) Population: all participants who gave informed consent, were randomised, and received at least one dose of double-blind study medication.Only participants who had assessment of the measure the day after double-blind treatment were analyzed.
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | Placebo | Eszopiclone | Zopiclone
Number analyzed (Participants) | 89 | 87 | 90
milliseconds
  7.5 hours post-dose, n=89, 87, 90 | 746.88 (10.36) | 791.99 (10.40) | 806.31 (10.33)
  8 hours post-dose, n=88, 87, 90 | 744.90 (10.44) | 787.41 (10.50) | 799.53 (10.40)
  8.5 hours post-dose, n=89, 87, 90 | 757.72 (10.44) | 793.18 (10.51) | 797.92 (10.39)
  9 hours post-dose, n=89, 87, 90 | 760.11 (10.75) | 802.53 (10.81) | 811.11 (10.69)
  9.5 hours post-dose, n=89, 87, 90 | 763.65 (10.17) | 793.69 (10.23) | 789.63 (10.13)
  10 hours post-dose, n=89, 87, 90 | 756.67 (10.54) | 778.09 (10.60) | 792.00 (10.48)
  10.5 hours post-dose, n=89, 87, 90 | 765.98 (10.55) | 774.06 (10.59) | 779.80 (10.51)
  11 hours post-dose, n=89, 87, 90 | 762.43 (9.88) | 760.29 (9.95) | 765.56 (9.85)
  11.5 hours post-dose, n=89, 87, 90 | 745.26 (9.48) | 750.79 (9.52) | 766.44 (9.44)

4. Secondary Outcome: Critical Flicker Fusion Test-Ascending Threshold
Description: Critical Flicker Fusion (CFF) is a validated cognitive assessment task that provides an index of central nervous system (CNS) activity and attention modulated motion detection. Participants are required to discriminate flicker from fusion, and vice versa, in a set of four light-emitting diodes arranged in a one-centimetre square. These diodes are held in foveal fixation when viewed at a distance of one metre. Individual thresholds are determined on four ascending and four descending scales. The mean of the four ascending presentations give the ascending threshold frequency in hertz.
Time Frame: 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: hertz
Arm/Group | Placebo | Eszopiclone | Zopiclone
Number analyzed (Participants) | 89 | 87 | 90
hertz
  7.5 hours post-dose, n=88, 87, 90 | 30.65 (0.24) | 30.84 (0.24) | 30.93 (0.24)
  8 hours post-dose, n=89, 87, 90 | 30.31 (0.24) | 30.30 (0.24) | 30.41 (0.24)
  8.5 hours post-dose, n=89, 87, 90 | 30.27 (0.22) | 29.98 (0.22) | 30.17 (0.22)
  9 hours post-dose, n=89, 87, 90 | 30.10 (0.23) | 29.90 (0.23) | 30.00 (0.23)
  9.5 hours post-dose, n=89, 87, 90 | 30.18 (0.23) | 29.99 (0.23) | 30.05 (0.23)
  10 hours post-dose, n=89, 87, 90 | 30.20 (0.24) | 29.91 (0.24) | 29.97 (0.23)
  10.5 hours post-dose, n=89, 87, 89 | 30.26 (0.21) | 29.99 (0.22) | 30.16 (0.21)
  11 hours post-dose, n=89, 87, 90 | 30.20 (0.23) | 30.06 (0.23) | 30.04 (0.23)
  11.5 hours post-dose, n=89, 87, 90 | 30.31 (0.22) | 30.28 (0.23) | 30.56 (0.22)

5. Secondary Outcome: Critical Flicker Fusion Test -Descending Threshold
Description: Analysis was performed on the individual assessments conducted at 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind) The mean of the four descending presentations from the CFF give the descending threshold frequency in hertz.
Time Frame: 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hertz
Arm/Group | Placebo | Eszopiclone | Zopiclone
Number analyzed (Participants) | 89 | 87 | 90
hertz
  7.5 hours post-dose, n=88, 87, 90 | 29.06 (0.35) | 28.37 (0.35) | 28.05 (0.35)
  8 hours post-dose, n=89, 87, 90 | 28.52 (0.33) | 27.95 (0.33) | 27.95 (0.33)
  8.5 hours post-dose, n=89, 87, 90 | 28.42 (0.34) | 27.75 (0.35) | 27.59 (0.34)
  9 hours post-dose, n=89, 87, 90 | 28.07 (0.34) | 27.64 (0.35) | 27.89 (0.34)
  9.5 hours post-dose, n=89, 87, 90 | 28.19 (0.34) | 27.81 (0.35) | 27.75 (0.34)
  10 hours post-dose, n=89, 87, 90 | 28.18 (0.34) | 27.96 (0.34) | 28.06 (0.34)
  10.5 hours post-dose, n=89, 87, 89 | 28.48 (0.34) | 27.99 (0.34) | 28.10 (0.34)
  11 hours post-dose, n=89, 87, 90 | 28.53 (0.34) | 28.03 (0.34) | 28.20 (0.34)
  11.5 hours post-dose, n=89, 87, 90 | 28.57 (0.33) | 28.69 (0.34) | 28.48 (0.33)

6. Secondary Outcome: Critical Flicker Fusion Test-Overall Threshold
Description: Analysis was performed on the individual assessments conducted at 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind) The mean of the four ascending and four descending presentations of the CFF give the overall threshold frequency in hertz.
Time Frame: 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: hertz
Arm/Group | Placebo | Eszopiclone | Zopiclone
Number analyzed (Participants) | 89 | 87 | 90
hertz
  7.5 hours post-dose, n=88, 87, 90 | 29.82 (0.26) | 29.57 (0.26) | 29.45 (0.26)
  8 hours post-dose, n=89, 87, 90 | 29.41 (0.25) | 29.11 (0.25) | 29.00 (0.24)
  8.5 hours post-dose, n=89, 87, 90 | 29.36 (0.25) | 28.86 (0.25) | 28.88 (0.25)
  9 hours post-dose, n=89, 87, 90 | 29.10 (0.25) | 28.79 (0.25) | 28.96 (0.25)
  9.5 hours post-dose, n=89, 87, 90 | 29.19 (0.25) | 28.90 (0.25) | 28.90 (0.25)
  10 hours post-dose, n=89, 87, 90 | 29.20 (0.25) | 28.95 (0.25) | 29.02 (0.25)
  10.5 hours post-dose, n=89, 87, 89 | 29.38 (0.24) | 29.00 (0.24) | 29.14 (0.24)
  11 hours post-dose, n=89, 87, 90 | 29.37 (0.25) | 29.07 (0.25) | 29.14 (0.25)
  11.5 hours post-dose, n=89, 87, 90 | 29.46 (0.24) | 29.50 (0.25) | 29.53 (0.24)

7. Secondary Outcome: Total Number of Attempted Symbol Substitutions, as Assessed by the Digit Symbol Substitution Test
Description: Analysis was performed on the individual assessments conducted at 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind). The Digit Symbol Substitution Test (DSST) is a pen and paper test that consists of rows of blank squares paired with randomly assigned digits (between 0 and 9). Participants are required to substitute each digit with a different nonsense symbol, according to a key printed at the top of the sheet that indicates the nonsense symbol that corresponds to each digit. Participants are given 120 seconds in which to complete the test.
Time Frame: 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: number of substitutions
Arm/Group | Placebo | Eszopiclone | Zopiclone
Number analyzed (Participants) | 89 | 87 | 90
number of substitutions
  7.5 hours post-dose, n=89, 87, 90 | 68.2 (1.09) | 64.7 (1.10) | 63.4 (1.09)
  8 hours post-dose, n=87, 84, 88 | 70.4 (1.16) | 66.5 (1.17) | 65.6 (1.15)
  8.5 hours post-dose, n=89, 87, 90 | 70.6 (1.13) | 67.4 (1.13) | 66.3 (1.12)
  9 hours post-dose, n=88, 87, 90 | 68.1 (1.20) | 65.2 (1.20) | 64.2 (1.19)
  9.5 hours post-dose, n=88, 87, 90 | 70.2 (1.12) | 67.2 (1.13) | 66.5 (1.12)
  10 hours post-dose, n=89, 87, 90 | 70.9 (1.14) | 68.2 (1.14) | 67.6 (1.13)
  10.5 hours post-dose, n=86, 85, 88 | 71.8 (1.16) | 69.7 (1.17) | 67.8 (1.16)
  11 hours post-dose, n=88, 87, 90 | 70.9 (1.11) | 68.1 (1.11) | 67.6 (1.10)
  11.5 hours post-dose, n=89, 87, 90 | 69.0 (1.16) | 68.0 (1.17) | 68.3 (1.16)

8. Secondary Outcome: Total Number of Correct Symbol Substitutions, as Assessed by the Digital Symbol Substitution Test
Description: as for outcome 7
Time Frame: 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: number of substitutions
Arm/Group | Placebo | Eszopiclone | Zopiclone
Number analyzed (Participants) | 89 | 87 | 90
number of substitutions
  7.5 hours post-dose, n=89, 87, 90 | 67.9 (1.10) | 64.3 (1.10) | 63.0 (1.10)
  8 hours post-dose, n=87, 84, 88 | 70.2 (1.16) | 66.2 (1.17) | 65.2 (1.16)
  8.5 hours post-dose, n=89, 87, 90 | 70.4 (1.13) | 67.0 (1.14) | 66.0 (1.13)
  9 hours post-dose, n=88, 87, 90 | 67.9 (1.20) | 64.8 (1.21) | 63.8 (1.20)
  9.5 hours post-dose, n=88, 87, 90 | 69.9 (1.12) | 66.9 (1.13) | 66.2 (1.12)
  10 hours post-dose, n=89, 87, 90 | 70.8 (1.14) | 68.0 (1.15) | 67.3 (1.14)
  10.5 hours post-dose, n=86, 85, 88 | 71.5 (1.17) | 69.5 (1.17) | 67.4 (1.16)
  11 hours post-dose, n=88, 87, 90 | 70.6 (1.11) | 67.8 (1.11) | 67.3 (1.10)
  11.5 hours post-dose, n=89, 87, 90 | 68.7 (1.16) | 67.8 (1.17) | 68.0 (1.12)

9. Secondary Outcome: 1-Back Percentage of Correct Responses
Description: The N-Back task requires the participant to indicate, using the mouse, whether the current stimulus presented on the screen and the one immediately before it visually match (i.e., "one-back"). In the versions of the tests used in this study, the stimuli are presented on screen for 500 ms, and the interval between stimuli is 2500 ms, with a ratio of 1:2 of "match" trials to non-match trials. The duration of the test is 2 minutes. The percentage of correct responses is the percentage of correct responses given in 2 minutes.
Time Frame: 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of responses
Arm/Group | Placebo | Eszopiclone | Zopiclone
Number analyzed (Participants) | 89 | 87 | 90
percentage of responses
  7.5 hours post-dose, n=87, 87, 88 | 93.9 (0.95) | 92.2 (0.96) | 90.4 (0.95)
  8 hours post-dose, n=89, 87, 89 | 93.3 (0.97) | 92.0 (0.98) | 89.5 (0.97)
  8.5 hours post-dose, n=89, 87, 90 | 93.6 (1.05) | 92.8 (1.06) | 89.6 (1.05)
  9 hours post-dose, n=89, 87, 90 | 93.5 (1.07) | 91.6 (1.08) | 89.4 (1.07)
  9.5 hours post-dose, n=89, 86, 90 | 92.9 (1.02) | 91.2 (1.02) | 90.7 (1.01)
  10 hours post-dose, n=89, 87, 90 | 93.0 (0.90) | 92.2 (0.91) | 92.0 (0.90)
  10.5 hours post-dose, n=89, 86, 89 | 94.4 (0.94) | 92.0 (0.95) | 91.7 (0.94)
  11 hours post-dose, n=89, 87, 90 | 93.0 (0.92) | 92.6 (0.93) | 91.9 (0.92)
  11.5 hours post-dose, n=89, 87, 90 | 93.4 (0.92) | 94.0 (0.92) | 92.0 (0.91)

10. Secondary Outcome: 3-Back Percentage of Correct Responses
Description: Analysis was performed on the individual assessments conducted at 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind). In "3-back" tasks, a comparison is made between the current stimulus and the two before the immediately preceding stimulus. In the versions of the tests used in this study, the stimuli are presented on screen for 500 ms, and the interval between stimuli is 2500 ms, with a ratio of 1:2 of "match" trials to non-match trials. The duration of the test is 2 min. The percentage of correct responses is the percentage of correct responses given in 2 min.
Time Frame: 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of responses
Arm/Group | Placebo | Eszopiclone | Zopiclone
Number analyzed (Participants) | 89 | 87 | 90
percentage of responses
  7.5 hours post-dose, n=87, 87, 88 | 84.6 (1.40) | 80.4 (1.41) | 76.9 (1.40)
  8 hours post-dose, n=89, 87, 89 | 83.5 (1.55) | 82.3 (1.56) | 76.8 (1.55)
  8.5 hours post-dose, n=89, 87, 90 | 82.4 (1.56) | 81.1 (1.57) | 78.3 (1.55)
  9 hours post-dose, n=89, 87, 90 | 83.3 (1.61) | 78.9 (1.62) | 77.3 (1.60)
  9.5 hours post-dose, n=89, 86, 90 | 82.1 (1.60) | 80.2 (1.61) | 76.9 (1.59)
  10 hours post-dose, n=89, 87, 90 | 83.4 (1.53) | 82.0 (1.54) | 79.2 (1.52)
  10.5 hours post-dose, n=89, 86, 89 | 82.6 (1.50) | 81.3 (1.51) | 79.7 (1.50)
  11 hours post-dose, n=89, 87, 90 | 81.7 (1.44) | 83.2 (1.45) | 79.8 (1.44)
  11.5 hours post-dose, n=89, 87, 90 | 82.9 (1.40) | 83.6 (1.41) | 81.1 (1.39)

11. Secondary Outcome: 1-Back Reaction Time
Description: Analysis was performed on the individual assessments conducted at 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind). Reaction time is the time taken to respond to a stimulus.
Time Frame: 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | Placebo | Eszopiclone | Zopiclone
Number analyzed (Participants) | 89 | 87 | 90
milliseconds
  7.5 hours post-dose, n=87, 87, 88 | 755.9 (17.81) | 819.3 (17.85) | 840.3 (17.75)
  8 hours post-dose, n=89, 87, 89 | 752.7 (16.89) | 783.7 (16.99) | 805.8 (16.87)
  8.5 hours post-dose, n=89, 87, 90 | 741.1 (17.09) | 776.1 (17.18) | 778.7 (17.04)
  9 hours post-dose, n=89, 87, 90 | 734.8 (16.58) | 784.5 (16.68) | 791.1 (16.58)
  9.5 hours post-dose, n=89, 86, 90 | 729.0 (16.84) | 757.2 (16.98) | 784.0 (16.80)
  10 hours post-dose, n=89, 87, 90 | 724.7 (16.39) | 760.8 (16.48) | 759.5 (16.34)
  10.5 hours post-dose, n=89, 86, 89 | 713.2 (15.81) | 735.2 (15.92) | 750.7 (15.80)
  11 hours post-dose, n=89, 87, 90 | 718.5 (16.26) | 716.9 (16.33) | 741.7 (16.22)
  11.5 hours post-dose, n=89, 87, 90 | 709.3 (16.83) | 716.7 (16.92) | 720.5 (16.78)

12. Secondary Outcome: 3-Back Reaction Time
Description: as for outcome 11
Time Frame: 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | Placebo | Eszopiclone | Zopiclone
Number analyzed (Participants) | 89 | 87 | 90
milliseconds
  7.5 hours post-dose, n=87, 87, 88 | 959.5 (20.87) | 1020.9 (20.87) | 1076.4 (20.79)
  8 hours post-dose, n=89, 87, 89 | 960.0 (21.56) | 1018.5 (21.62) | 1042.2 (21.53)
  8.5 hours post-dose, n=89, 87, 90 | 925.9 (21.37) | 997.7 (21.49) | 1024.2 (21.33)
  9 hours post-dose, n=89, 87, 90 | 916.9 (21.50) | 1002.2 (21.61) | 1007.8 (21.46)
  9.5 hours post-dose, n=89, 86, 90 | 932.9 (21.86) | 992.1 (22.05) | 978.0 (21.81)
  10 hours post-dose, n=89, 87, 90 | 907.4 (21.26) | 948.7 (21.36) | 987.5 (21.19)
  10.5 hours post-dose, n=89, 86, 89 | 900.3 (20.92) | 961.5 (21.08) | 945.2 (20.89)
  11 hours post-dose, n=89, 87, 90 | 915.3 (19.61) | 935.5 (19.70) | 940.4 (19.54)
  11.5 hours post-dose, n=89, 87, 90 | 876.2 (20.49) | 903.2 (20.58) | 934.7 (20.39)

13. Secondary Outcome: Sedation Score, as Assessed by the Linear Analogue Rating Scales
Description: The Linear Analogue Rating Scale (LARS) is used as a measure of the subjective effects of psychoactive drugs. Participants mark a series of 10 cm (100 unit line) analogue scales (1-100, 100 = most impaired) relating to dizzy, clumsy, anxious, relaxed, tired, drowsy, alert, energetic, sad, and depressed, indicating their present feeling with regard to a mid-point, representing their "usual" state of mind before treatment began. The higher the score, the more impaired the participant feels. The Tiredness, Alertness, Energy, and Drowsiness scores are averaged to derive an overall Sedation score.
Time Frame: 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | Eszopiclone | Zopiclone
Number analyzed (Participants) | 89 | 87 | 90
points on a scale
  7.5 hours post-dose, n=89, 87, 90 | 54.21 (1.15) | 54.87 (1.16) | 57.00 (1.14)
  8 hours post-dose, n=89, 87, 90 | 54.54 (1.37) | 56.40 (1.15) | 59.21 (1.13)
  8.5 hours post-dose, n=89, 87, 90 | 54.07 (1.18) | 54.39 (1.19) | 56.93 (1.18)
  9 hours post-dose, n=89, 87, 90 | 53.63 (1.12) | 54.93 (1.12) | 56.01 (1.10)
  9.5 hours post-dose, n=89, 87, 90 | 53.84 (1.14) | 55.39 (1.15) | 55.90 (1.13)
  10 hours post-dose, n=89, 87, 90 | 53.98 (1.21) | 54.68 (1.23) | 55.73 (1.21)
  10.5 hours post-dose, n=89, 87, 90 | 51.77 (1.21) | 53.77 (1.13) | 55.31 (1.12)
  11 hours post-dose, n=89, 87, 90 | 51.47 (1.06) | 51.49 (1.06) | 52.79 (1.05)
  11.5 hours post-dose, n=89, 87, 90 | 49.02 (1.21) | 49.41 (1.22) | 51.24 (1.20)

14. Secondary Outcome: Mood Score, as Assessed by the Linear Analogue Rating Scales
Description: Analysis was performed on the individual assessments conducted at 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind). The Anxiety, Depression, Relaxed, and Sadness scores are averaged to derive an overall "Mood" score (as described in Outcome Measure 14). Each item was assessed on a 1-100 point scale, where 100 indicates most impaired.
Time Frame: 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | Eszopiclone | Zopiclone
Number analyzed (Participants) | 89 | 87 | 90
points on a scale
  7.5 hours post-dose, n=89, 87, 90 | 47.75 (0.71) | 48.13 (0.72) | 48.03 (0.71)
  8 hours post-dose, n=89, 87, 90 | 49.19 (0.71) | 48.42 (0.71) | 49.11 (0.70)
  8.5 hours post-dose, n=89, 87, 90 | 48.88 (0.70) | 48.42 (0.70) | 48.30 (0.69)
  9 hours post-dose, n=89, 87, 90 | 48.48 (0.74) | 47.67 (0.75) | 48.61 (0.74)
  9.5 hours post-dose, n=89, 87, 90 | 48.30 (0.75) | 47.89 (0.76) | 47.54 (0.75)
  10 hours post-dose, n=89, 87, 90 | 47.98 (0.79) | 48.25 (0.79) | 48.28 (0.78)
  10.5 hours post-dose, n=89, 87, 90 | 47.57 (0.87) | 48.72 (0.88) | 48.47 (0.87)
  11 hours post-dose, n=89, 87, 90 | 47.45 (0.85) | 47.07 (0.86) | 47.90 (0.85)
  11.5 hours post-dose, n=89, 87, 90 | 45.63 (1.03) | 47.09 (1.40) | 46.08 (1.03)

15. Secondary Outcome: Coordination Score, as Assessed by the Linear Analogue Rating Scales
Description: Analysis was performed on the individual assessments conducted at 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind). The Dizziness and Clumsiness scores are averaged to derive an overall "Coordination" score (as described in Outcome Measure 14). Each item was assessed on a 1-100 point scale, where 100 indicates most impaired.
Time Frame: 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, and 11.5 hours post-dose (double-blind)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | Eszopiclone | Zopiclone
Number analyzed (Participants) | 89 | 87 | 90
points on a scale
  7.5 hours post-dose, n=89, 87, 90 | 49.09 (1.13) | 50.33 (1.15) | 52.42 (1.13)
  8 hours post-dose, n=89, 87, 90 | 50.03 (0.92) | 51.21 (0.93) | 52.10 (0.92)
  8.5 hours post-dose, n=89, 87, 90 | 49.23 (0.86) | 49.52 (0.87) | 51.76 (0.86)
  9 hours post-dose, n=89, 87, 90 | 49.68 (0.94) | 50.38 (0.95) | 50.41 (0.94)
  9.5 hours post-dose, n=89, 87, 90 | 49.08 (0.97) | 49.42 (0.98) | 51.41 (0.96)
  10 hours post-dose, n=89, 87, 90 | 49.37 (0.96) | 49.72 (0.97) | 50.27 (0.95)
  10.5 hours post-dose, n=89, 87, 90 | 48.60 (0.86) | 50.68 (0.87) | 50.40 (0.86)
  11 hours post-dose, n=89, 87, 90 | 48.97 (0.83) | 48.51 (0.84) | 49.96 (0.83)
  11.5 hours post-dose, n=89, 87, 90 | 48.20 (0.82) | 47.45 (0.83) | 49.82 (0.81)

ADVERSE EVENTS:
Arm/Group | Placebo | Eszopiclone | Zopiclone
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/88 | 0/90
Other Adverse Events (participants affected / at risk) | 12/89 | 44/88 | 44/90
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=89) | Eszopiclone (N=88) | Zopiclone (N=90)
Dysgeusia (Nervous system disorders) | 0 | 27 | 30
Somnolence (Nervous system disorders) | 1 | 11 | 7
Dizziness (Nervous system disorders) | 0 | 4 | 5
Headache (Nervous system disorders) | 2 | 2 | 2
Disturbance in attention (Nervous system disorders) | 0 | 2 | 3
Paraesthesia (Nervous system disorders) | 1 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 1
Coordination abnormal (Nervous system disorders) | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 1
Poor quality sleep (Nervous system disorders) | 0 | 1 | 0
Fatigue (General disorders) | 4 | 6 | 6
Asthenia (General disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 2 | 0
Nightmare (Psychiatric disorders) | 0 | 2 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0
Fear (Psychiatric disorders) | 0 | 1 | 0
Somnambulism (Psychiatric disorders) | 0 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 1 | 1
Eye pruritis (Eye disorders) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.